CLINICAL TRIAL: NCT03813511
Title: Prevalence and Dynamics of Sleep-Disordered Breathing (SDB) in Patients With Severe Valvular Regurgitation and High Surgical Risk Undergoing Minimally Invasive Clip Procedure
Brief Title: Sleep-Disordered Breathing in Patients With Severe Valvular Regurgitation Undergoing Clip Procedure
Acronym: ClipSDB
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Principal Investigator, Muhammed Gerçek, Principal Investigator, Heart and Diabetes Center North-Rhine Westfalia
Other Study IDs: HDZ-KA_015_MG
Record Dates: First submitted 2018-12-19; First posted 2019-01-23 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Sleep Disordered Breathing; Valvular Regurgitation
Keywords: Minimally invasive surgery; Clip procedure
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In a prospective observational study, the investigators investigate the prevalence of sleep disordered breathing in patients with severe valvular regurgitation and the effect of using the minimal invasive Clip technique on sleep disordered breathing.

DETAILED DESCRIPTION:
The purpose of this study is to analyze the prevalance of sleep disordered breathing in patients with severe valvular regurgitation and the impact of a therapy with the minimal-invasive Clip technique.

Therefore, the investigators want to include consecutive patients with unknown sleep-associated respiratory distress syndrome and, in addition, as a study-specific achievement, the investigators want to obtain the quality of life and specific symptoms of the patients by using established questionnaires. After three month of post-interventional care, the patients will get a post-interventional check-up in our cardiological outpatient clinic, where the course of sleep-associated respiratory distress syndrome and the actual quality of life and specific symptoms will be documented by using a cardiorespiratory polygraphy and the same questionnaires.

The entire hospital stay, including possible post-interventional complications, will be documented for this study from the patients' medical records. The routine examinations (laboratory values, ECG, 6-minute walk test, pulmonary function examinations, spiroergometry, transthoracic / -oesophageal echocardiography, etc.) shall also be recorded in the database of this study.

The plan is to include 100 evaluable patients with complete follow-up and the associated test results. For this purpose, a screening of 150 patients is expected to be required.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe valvular regurgitation and currently unknown sleep disorder breathing who will be treated with a minimal invasive Clip technique

Exclusion Criteria:

* Patients with more then one valvular disease which requires Treatment
* Patients with complex congenital heart disease
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stationäre patients with severe valvular regurgitation and currently unknown sleep disorder breathing who will be treated with a minimal invasive Clip technique
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalance of Sleep disordered breathing in Patiens with severe valvular regurgitation | 3 month
  Proportion of of Sleep disordered breathing in Patiens with severe valvular regurgitation in a given time period
Influence of the minimal invasive Clip technique on apnea-hypopnea index | 3 month
  Changes on the number of apnea and hypopnea events per hour of sleep due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on apnea index | 3 month
  Changes on the number of apnea events per hour of sleep due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on the oxygen desaturation index | 3 month
  Changes on the number of times per hour of sleep that the blood's oxygen level drop by a certain degree from baseline due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on T90 | 3 month
  Changes on the the percentage of time during which arterial O2 saturation was less than 90% (T90) due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on sleep cycle length | 3 month
  Changes on the duration of the five stages of sleep (in minutes) due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on ventilation length during sleep | 3 month
  Changes on the ventilation length (in seconds) due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on PISA in tranthoracic echocardiography | 3 month
  Changes on the proximal isovelocity hemispheric surface area (PISA in square millimeter) in tranthoracic echocardiography due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on the effective regurgitant orifice (ERO) in tranthoracic echocardiography | 3 month
  Changes on the effective regurgitant orifice (ERO in square millimeter) in tranthoracic echocardiography due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on the peak velocity of the mitral regurgitant jet (mR-Vmax) in tranthoracic echocardiography | 3 month
  Changes on the peak velocity of the mitral regurgitant jet (mR-Vmax in meter per seconds) in tranthoracic echocardiography due to the minimal invasiv Clip technique
Influence of the minimal invasive Clip technique on the myocardial perfomance index (TEI-index) in tranthoracic echocardiography | 3 month
  Changes on systolic and diastolic time intervals in expressing global systolic and diastolic ventricular function (without unity) in tranthoracic echocardiography due to the minimal invasiv Clip technique

SECONDARY OUTCOMES:
Post-interventional changes in daytime sleepiness with and without sleep disordered breathing | 3 month
  Post-interventional changes in daytime sleepiness with and without sleep disordered breathing measured by the Epworth Sleepinss Scale (ESS) (From 0 to 24 point-scale; A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates severe daytime sleepiness)
Post-interventional survey of patient health with and without sleep disordered breathing | 3 month
  Post-interventional survey of patient health with and without sleep disordered breathing measured by the Short Form (36) Health Survey (SF-36).
  SF-36 consists of eight scaled score (Vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health). Total range from 0 to 100 points (from worst to best)
Post-interventional assesment of Symptoms, function and quallity of life with and without sleep disordered breathing by patients with heart failure | 3 month
  Post-interventional assesment of Symptoms, function and quallity of life with and without sleep disordered breathing by patients with heart failure using the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) that hat quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Total range is from 0 to 100 points. 0 denotes the worst and 100 the best possible health status
Post-interventional measurement of the adverse effects of heart failure on patient's life with and without sleep disordered breathing | 3 month
  Post-interventional measurement of the adverse effects of heart failure on patient's life with and without sleep disordered breathing using the Minnesota Living with Heart Failure Questionnaire. It provides a total score range 0-105, from best to worst
Post-interventional assessment of the sleep quality with and without sleep disordered breathing | 3 month
  Post-interventional assessment of the sleep quality with and without sleep disordered breathing using the Pittsburgh Sleep Quality Index (PSQI) (From 0 (worst) to 21 (best))
Post-interventional changes in generic health status. with and without sleep disordered breathing | 3 month
  Post-interventional changes in generic health status. with and without sleep disordered breathing using the EQ-5D questionnaire (grade ranging from 0, the worst possible health status, to 100 ,the best possible health status
Post-interventional changes aerobic capacity and endurance with and without sleep disordered breathing | 3 month
  Post-interventional changes on aerobic capacity and endurance with and without sleep disordered breathing using the cardiopulmonary exercise testing (vO2max in milliliter per minute per kilogram
Post-interventional changes functional capacity of cardiopulmonary and musculoskeletal system with and without sleep disordered breathing | 3 month
  Post-interventional changes on aerobic capacity and endurance with and without sleep disordered breathing using the six minutes walk test (in meters)
Post-interventional changes on cognitive functions with and without sleep disordered breathing | 3 month
  Post-interventional changes on cognitive functions with and without sleep disordered breathing using the Montreal Cognitive Assessment Test (MOCA) (From 0 (worst) to 30 (best) point-scale)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Gercek, MD, Principal Investigator — Heart and Diabetes Center North Rhine-Westphalia
Locations (1):
- Herz- und Diabeteszentrum NRW, Ruhr-Universität Bochum, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No